CLINICAL TRIAL: NCT06016504
Title: Development and Evaluation of an Adaptive Virtual Consultation Tool for Prostate Cancer Patients
Brief Title: Adaptive Virtual Consultation Tool to Enhance Education and Understanding in Patients with Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low/slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mitchell Humphreys, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-002955; NCI-2022-09812 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-002955 (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2023-08-01; First posted 2023-08-29 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (AVCT) (Experimental): Patients participate in an adaptive virtual consultation on trial.
  Interventions: Behavioral: Health Education; Other: Survey Administration
- Arm 2 (non-AVCT) (Active Comparator): Patients participate in a non-adaptive virtual consultation on trial.
  Interventions: Behavioral: Health Education; Other: Survey Administration
- Arm 3 (information-only) (Active Comparator): Patients receive information-only on trial.
  Interventions: Other: Informational Intervention; Other: Survey Administration

INTERVENTIONS:
Behavioral: Health Education — Participate in an adaptive virtual consultation
  Arms: Arm 1 (AVCT)
Behavioral: Health Education — Participate in a non-adaptive virtual consultation
  Arms: Arm 2 (non-AVCT)
Other: Informational Intervention — Given information-only
  Arms: Arm 3 (information-only)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial aims to design and validate an adaptive virtual consultation tool (AVCT) for men with prostate cancer (PC). An AVCT utilizes health literacy assessments in combination with learning preferences and individual disease characteristics to provide focused and guided knowledge on PC tailored to the individual patient. Using an AVCT to enhance patient education may improve patient understanding and result in higher patient satisfaction with treatment decisions amongst men with PC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop an adaptive virtual consultation tool for PC (AVCT):

Ia. To incorporate and integrate the inputs from a diverse group of patients (including minorities), patient advocates, nursing, physicians and education experts in the design process for the adaptive consultation tool; Ib. Employ user centered iterative design approach to develop an adaptive learning tool on mobile devices that is tailored to individuals based on symptoms, health literacy, learning style, and disease specific characteristics.

II. To assess the feasibility, acceptability and usability of AVCT:

IIa. To validate the design approach and customization rules at the completion of the participatory design process using a convenience sample of subjects through assessment of system interaction logs and qualitative feedback from users on cognition, ease-of-use, usability and customization efficacy; IIb. To utilize the feasibility study results in (2a) to refine the interface, information presentation, and adaptive customization approach.

III. To determine the efficacy of AVCT using a small-scale comparative study:

IIIa. To design and execute a three arm comparative study consisting of adaptive virtual consultation, non-adaptive virtual consultation and standard-practice information-only control intervention and assess the comparative efficacy of the tool on the main outcome variable, satisfaction with health care episode; IIIb. To measure changes in other outcome variables at baseline, post-intervention, 3-month and 12-month duration; IIIc. To analyze the mediating influence of decision self-efficacy and a number of moderating factors including preference for decision-making participation and health literacy on outcome variables.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM 1: Patients participate in an adaptive virtual consultation on trial.

ARM 2: Patients participate in a non-adaptive virtual consultation on trial.

ARM 3: Patients receive information-only on trial.

After completion of study intervention, patients are followed up at 3- and 12-months post treatment decision.

ELIGIBILITY:
Inclusion Criteria:

* The participants in this study will be community dwelling, males with prostate cancer (PC) and their healthcare advocate, if applicable
* Proficiency in English is required

Exclusion Criteria:

* Mental incompetency to participate in the study and/or no treatment option due to other health reasons

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 18 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction measured by post utilization surveys | 3-month post treatment decision
  Patient's satisfaction is to be measured by post utilization surveys using general Likert scale assessment tools.
  Descriptive statistics will be used to summarize the data at each study time point. For all the measures collected at multiple time points, generalized linear equations (GEE) will be used to evaluate the effect of treatment and time adjusting for usage pattern.
Patient satisfaction measured by post utilization surveys | 12-month post treatment decision
  Patient's satisfaction is to be measured by post utilization surveys using general Likert scale assessment tools.
  Descriptive statistics will be used to summarize the data at each study time point. For all the measures collected at multiple time points, generalized linear equations (GEE) will be used to evaluate the effect of treatment and time adjusting for usage pattern.
Health outcomes for cancer recurrence using PSA | Baseline
  Measured by Prostate specific antigen ( PSA )
Health outcomes for urinary function using IPSS | Baseline
  Measured using International Prostate symptom score (IPSS)
Health outcomes for sexual function using SHIM score | Baseline
  Measured using Sexual Health inventory for men (SHIM) score
Health outcomes for cancer recurrence using PSA | 3-month post treatment decision
  Measured by Prostate specific antigen ( PSA )
Health outcomes for urinary function | 3-month post treatment decision
  Measured using International Prostate symptom score (IPSS)
Health outcomes for sexual function | 3-month post treatment decision
  Measured using Sexual Health inventory for men (SHIM) score
Health outcomes for cancer recurrence using PSA | 12-months post treatment decision
  Measured by Prostate specific antigen ( PSA )
Health outcomes for urinary function | 12-months post treatment decision
  Measured using International Prostate symptom score (IPSS)
Health outcomes for sexual function | 12-months post treatment decision
  Measured using Sexual Health inventory for men (SHIM) score

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell R. Humphreys, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials